CLINICAL TRIAL: NCT04519697
Title: A Phase IB/IIA Study of Adult Allogeneic Bone Marrow Derived Mesenchymal Stem Cells for the Treatment of Rectovaginal Fistulas in the Setting of Crohn's Disease.
Brief Title: Mesenchymal Stem Cells for the Treatment of Rectovaginal Fistulas in Participants With Crohn's Disease
Acronym: RVF
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amy Lightner (Other)
Responsible Party: Sponsor-Investigator, Amy Lightner, Sponsor-investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 20-936
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Rectovaginal Fistula; Crohn Disease; Crohn Disease of Vulva; Rectolabial; Fistula
Keywords: Crohn's disease; rectovaginal fistula; mesenchymal stem cells; mesenchymal stem cell
MeSH Terms: conditions — Rectovaginal Fistula; Crohn Disease; Fistula

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mesenchymal Stem Cells (Experimental): Direct injection of adult allogeneic bone marrow derived mesenchymal stem cells at a dose of 75 million cells into rectovaginal fistula at baseline with a possible repeat injection at 3 months if not completely healed from the first injection.
  Interventions: Drug: Mesenchymal Stem Cells
- Placebo (Placebo Comparator): Direct injection of normal saline with a possible repeat injection at 3 months if not completely healed from the first injection. If not completely healed after 6 months, participants will then cross over to the treatment group to receive a direct injection of adult allogeneic bone marrow derived mesenchymal stem cells at a dose of 75 million cells into rectovaginal fistula.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mesenchymal Stem Cells — Adult allogeneic bone marrow derived mesenchymal stem cells for the treatment of rectovaginal fistulas in the setting of Crohn's disease.
  Arms: Mesenchymal Stem Cells
Other: Placebo — Normal Saline
  Arms: Placebo

SUMMARY:
Approximately 10% of all female Crohn's patients have a rectovaginal fistula. Rectovaginal fistulas cause air, stool, and/or drainage per vagina and may be associated with pain, recurrent urinary tract infections and diminished quality of life. Conventional therapy includes immunosuppressive medications used to treat Crohn's disease and various surgical interventions. However, all have limited ability to heal these fistulas. The purpose of this study is to determine the safety and efficacy of using allogeneic bone marrow derived mesenchymal stem cells (MSCs) to treat people with rectovaginal fistulas in the setting of Crohn's disease.

DETAILED DESCRIPTION:
This study is designed to determine the safety and efficacy of direct injection of adult allogeneic bone marrow derived mesenchymal stem cells for the treatment of rectovaginal fistulas in the setting of Crohn's disease. The study will randomize 20 participants. Enrolled participants will be randomized to treatment group with MSCs versus placebo in a 3:1 fashion. Participants in the treatment group will have a direct injection of MSCs at a dose of 75 million cells. This will be given as a direct injection in and around the fistula tract. Participants will be evaluated for complete healing at three months. If complete healing has been achieved patients will continue to be followed for one year. If complete healing has not been achieved at three months, participants will be eligible for a second injection of MSCs at the same dose of 75 million cells. Control participants without complete healing from placebo will cross over at the six month visit to receive an injection of MSCs, and will be followed for one year after treatment for a total duration of 18 months.

ELIGIBILITY:
Inclusion Criteria:

1. Females 18-75 years of age with a diagnosis of Crohn's disease for at least six months duration.
2. Single-tract, rectovaginal fistula in the setting of Crohn's disease.
3. Have no contraindications to MR evaluations: e.g. pacemaker or magnetically active metal fragments, claustrophobia
4. Ability to comply with protocol
5. Competent and able to provide written informed consent, and ability to comply with protocol
6. Concurrent Crohn's related therapies with stable doses (>2 months) corticosteroids, 5-ASA drugs, immunomodulators, anti-TNF therapy, anti-integrin and anti-interleukin are permitted

Exclusion Criteria:

1. Inability to give informed consent.
2. Clinically significant medical conditions within the six months before administration of MSCs: e.g. myocardial infarction, active angina, congestive heart failure or other conditions that would, in the opinion of the investigators, compromise the safety of the subject.
3. Specific exclusions:

   1. Hepatitis B or C
   2. HIV
   3. Abnormal AST or ALT at screening(defined as >/= 2x ULN)
4. History of cancer including melanoma (with the exception of localized skin cancers) within one year of screening.
5. History of colorectal cancer within 5 years.
6. Investigational drug within 30 days of treatment
7. Pregnant or breast feeding or trying to become pregnant.
8. Presence of a rectovaginal or perineal body fistula
9. Change in Crohn's immunosuppressive regimen within the 2 months prior to enrollment
10. Uncontrolled intestinal Crohn's disease which will require escalation for medical therapy or surgery within 2 months of enrollment
11. Severe anal canal disease that is stenotic and requires dilation
12. Inability to wean corticosteroids
13. Unwilling to agree to use acceptable contraception methods during participation in study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2020-10-28 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Treatment related adverse events | Month 6
  Number of participants with treatment related adverse events post-injection of 75 million allogeneic bone marrow derived MSC's for the treatment of rectovaginal fistula in the setting of Crohn's disease as assessed by protocol CCF-Stem Cells IBD-003

SECONDARY OUTCOMES:
Complete clinical healing | Month 6, Month 12
  Number of participants with complete clinical healing post-injection of 75 million allogeneic bone marrow derived MSC's for the treatment of rectovaginal fistula in the setting of Crohn's disease.
  Complete healing is defined as:
  Radiographic Healing: MRI with an absence of a fluid collection >2 cm in 3 of 3 dimensions, lack of edema, inflammation or sign of active inflammatory response. A remnant scar of a fistula tract may remain
  Clinical Healing: 100% cessation of drainage on both clinical exam with deep palpation and per patient report and complete closure of the fistula tract upon assessment with an examination under anesthesia
Partial healing | Month 6, Month 12
  Number of participants with partial clinical healing post-injection of 75 million allogeneic bone marrow derived MSC's for the treatment of rectovaginal fistula in the setting of Crohn's disease
  Partial healing is defined as:
  Radiographic healing: MRI with an absence of a fluid collection >2 cm in 2 of 3 dimensions, lack of edema, inflammation or sign of active inflammatory response. A remnant scar of a fistula tract may remain
  Clinical healing: Greater than or equal to 50% cessation of drainage on both clinical exam with deep palpation and per patient report and partial closure of the fistula tract upon assessment with an examination under anesthesia
Lack of response | Month 6, Month 12
  Number of participants with lack of response post-injection of 75 million allogeneic bone marrow derived MSC's for the treatment of rectovaginal fistula in the setting of Crohn's disease
  Lack of Response is defined as: Radiographic and clinical healing which does not meet the threshold for Partial Healing
Worsening disease | Month 6, Month 12
  Number of participants with worsening disease post-injection of 75 million allogeneic bone marrow derived MSC's for the treatment of rectovaginal fistula in the setting of Crohn's disease
  Worsening disease is defined as:
  Radiographic: MRI with a fluid collection >2 cm in 2 of 3 dimensions, edema, inflammation or sign of active inflammatory response. An increased number of tracts may be seen, or increased branching from the primary tract,
  Clinical: Increased drainage per patient report and on clinical exam

CONTACTS AND LOCATIONS:
Overall Officials: Amy Lightner, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Background] Peyrin-Biroulet L, Loftus EV Jr, Colombel JF, Sandborn WJ. The natural history of adult Crohn's disease in population-based cohorts. Am J Gastroenterol. 2010 Feb;105(2):289-97. doi: 10.1038/ajg.2009.579. Epub 2009 Oct 27. PMID 19861953
- [Background] Schwartz DA, Loftus EV Jr, Tremaine WJ, Panaccione R, Harmsen WS, Zinsmeister AR, Sandborn WJ. The natural history of fistulizing Crohn's disease in Olmsted County, Minnesota. Gastroenterology. 2002 Apr;122(4):875-80. doi: 10.1053/gast.2002.32362. PMID 11910338
- [Background] Hannaway CD, Hull TL. Current considerations in the management of rectovaginal fistula from Crohn's disease. Colorectal Dis. 2008 Oct;10(8):747-55; discussion 755-6. doi: 10.1111/j.1463-1318.2008.01552.x. Epub 2008 May 4. PMID 18462243
- [Background] Panes J, Garcia-Olmo D, Van Assche G, Colombel JF, Reinisch W, Baumgart DC, Dignass A, Nachury M, Ferrante M, Kazemi-Shirazi L, Grimaud JC, de la Portilla F, Goldin E, Richard MP, Leselbaum A, Danese S; ADMIRE CD Study Group Collaborators. Expanded allogeneic adipose-derived mesenchymal stem cells (Cx601) for complex perianal fistulas in Crohn's disease: a phase 3 randomised, double-blind controlled trial. Lancet. 2016 Sep 24;388(10051):1281-90. doi: 10.1016/S0140-6736(16)31203-X. Epub 2016 Jul 29. PMID 27477896
- [Background] Panes J, Garcia-Olmo D, Van Assche G, Colombel JF, Reinisch W, Baumgart DC, Dignass A, Nachury M, Ferrante M, Kazemi-Shirazi L, Grimaud JC, de la Portilla F, Goldin E, Richard MP, Diez MC, Tagarro I, Leselbaum A, Danese S; ADMIRE CD Study Group Collaborators. Long-term Efficacy and Safety of Stem Cell Therapy (Cx601) for Complex Perianal Fistulas in Patients With Crohn's Disease. Gastroenterology. 2018 Apr;154(5):1334-1342.e4. doi: 10.1053/j.gastro.2017.12.020. Epub 2017 Dec 24. PMID 29277560
- [Background] Lightner AL, Dozois EJ, Dietz AB, Fletcher JG, Friton J, Butler G, Faubion WA. Matrix-Delivered Autologous Mesenchymal Stem Cell Therapy for Refractory Rectovaginal Crohn's Fistulas. Inflamm Bowel Dis. 2020 Apr 11;26(5):670-677. doi: 10.1093/ibd/izz215. PMID 31605115
- [Background] Garcia-Arranz M, Herreros MD, Gonzalez-Gomez C, de la Quintana P, Guadalajara H, Georgiev-Hristov T, Trebol J, Garcia-Olmo D. Treatment of Crohn's-Related Rectovaginal Fistula With Allogeneic Expanded-Adipose Derived Stem Cells: A Phase I-IIa Clinical Trial. Stem Cells Transl Med. 2016 Nov;5(11):1441-1446. doi: 10.5966/sctm.2015-0356. Epub 2016 Jul 13. PMID 27412883
- [Background] Sanz-Baro R, Garcia-Arranz M, Guadalajara H, de la Quintana P, Herreros MD, Garcia-Olmo D. First-in-Human Case Study: Pregnancy in Women With Crohn's Perianal Fistula Treated With Adipose-Derived Stem Cells: A Safety Study. Stem Cells Transl Med. 2015 Jun;4(6):598-602. doi: 10.5966/sctm.2014-0255. Epub 2015 Apr 29. PMID 25925838